CLINICAL TRIAL: NCT05545111
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of NBI-1117568 in Adults With Schizophrenia Who Warrant Inpatient Hospitalization
Brief Title: Efficacy, Safety, Tolerability, and Pharmacokinetics of NBI-1117568 in Adults With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1117568-SCZ2028
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; NBI-1117568; muscarinic
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level A (Experimental): Participant administered Dose Level A (6 weeks)
  Interventions: Drug: NBI-1117568
- Dose Level B (Experimental): Participant administered Dose Level B (6 weeks)
  Interventions: Drug: NBI-1117568
- Dose Level C (Experimental): Participant administered Dose Level C (6 weeks)
  Interventions: Drug: NBI-1117568
- Dose Level D (Experimental): Participant administered Dose Level D (6 weeks)
  Interventions: Drug: NBI-1117568
- Placebo Schedule (Placebo Comparator): Participant administered placebo (6 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-1117568 — Active treatment with orally administered NBI-1117568
  Arms: Dose Level A; Dose Level B; Dose Level C; Dose Level D
Drug: Placebo — Placebo matching NBI-1117568
  Arms: Placebo Schedule

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, multi-arm, multi-stage inpatient study designed to assess the efficacy, safety, tolerability, and pharmacokinetics (PK) of NBI-1117568 compared with placebo in adult subjects with a primary diagnosis of schizophrenia, who are experiencing an acute exacerbation or relapse of symptoms.

ELIGIBILITY:
Key Inclusion Criteria:

* Completed informed consent.
* Subject has a primary diagnosis of schizophrenia.
* The subject is experiencing an acute exacerbation or relapse of symptoms and currently requires hospitalization.
* Subjects taking prohibited medications, including antipsychotics, must discontinue before study participation
* Subject is willing and able to remain in an inpatient setting for the study duration, follow instructions, and comply with the protocol requirements.

Key Exclusion Criteria:

* An unstable medical condition, chronic disease, or malignancy.
* Considered by the investigator to be at imminent risk of suicide or injury to self or others.
* Diagnosis of moderate or severe substance use disorder (with the exception of nicotine or caffeine dependence) within 6 months prior to screening.
* Positive alcohol test or drug screen for disallowed substances.
* Have a history of poor or suspected poor compliance in clinical research studies and/or in the investigator's opinion, the subject is not capable of adhering to the protocol requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total Positive and Negative Syndrome Scale (PANSS) score at Week 6 | Baseline and Week 6
  The PANSS evaluates the severity of various symptoms of schizophrenia, and is commonly used to measure symptom reduction in patients taking antipsychotics. Each item is scored on a 7-point severity scale (1=absent; 2=minimal; 3=mild; 4=moderate; 5=moderate severe; 6=severe; 7=extreme). The PANSS total score is derived from the summation of each item. A higher score indicates greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (15):
- United States (15):
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, Rogers, Arkansas
  - Neurocrine Clinical Site, Lemon Grove, California
  - Neurocrine Clinical Site, Pico Rivera, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Torrance, California
  - Neurocrine Clinical Site, Miami Lakes, Florida
  - Neurocrine Clinical Site, Oakland Park, Florida
  - Neurocrine Clinical Site, Gaithersburg, Maryland
  - Neurocrine Clinical site, St Louis, Missouri
  - Neurocrine Clinical Site, Berlin, New Jersey
  - Neurocrine Clinical Site, North Canton, Ohio
  - Neurocrine Clinical Site, Austin, Texas
  - Neurocrine Clinical Site, DeSoto, Texas
  - Neurocrine Clinical Site, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No